CLINICAL TRIAL: NCT04502303
Title: A Prospective Study to Evaluate the Inflammation and Fibrosis of Intestinal Stricture in Patients With Crohn's Disease by 18F-FDG and 68Ga-FAPI PET/CT
Brief Title: 18F-FDG and 68Ga-FAPI PET/CT in Crohn's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAPICD
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: Patients with intestinal stricture will undergo 18F-FDG and 68Ga-FAPI PET/CT on two consecutive days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Crohn's disease: patients with intestinal stricture (Experimental): Patients with intestinal strictures confirmed by other modalities, e.g. CT, MR, ultrasound, and endoscopy, will be recruited in the study.
  Interventions: Diagnostic Test: 18F-FDG and 68Ga-FAPI PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-FDG and 68Ga-FAPI PET/CT — Participants will undergo 18F-FDG (0.12-0.15mCi/kg) and 68Ga-FAPI (3-6mCi) PET/CT on two consecutive days. At least 6 hours of fast is required for 18F-FDG PET scan, while no dietary control is necessary for 68Ga-FAPI PET scan. If the patients are on metformin, discontinuation of 48 hours is required before 18F-FDG injection to minimize the bowel uptake. If the patient is planned for surgical resection of one or more stricture (s), the scans have to be completed within a maximum period of 30 days before the surgery.

SUMMARY:
Intestinal stricture is a complication of Crohn's disease (CD), which is thought to be the result of chronic transmural inflammation combined with a dysregulated wound-healing process. While inflammatory strictures may respond to anti-inflammatory treatment, fibrotic strictures are usually anti-inflammation resistant, requiring further endoscopic balloon dilation or surgical intervention. Therefore, to determinate the inflammatory or fibrotic nature of intestinal stricture is a key step in the treatment of CD. 18F-FDG is a radiotracer reflecting the glucose metabolism of disease and is usually accumulated in inflammatory disease. 68Ga-FAPI is a novel radiotracer that specifically targets fibroblast activation protein (FAP). FAP is a membrane glycoprotein expressed on activated fibroblasts, which are key cells in the process of fibrotic intestinal stricture of CD. In this study, we hypothesis that the inflammatory or fibrotic nature of intestinal stricture can be non-invasively evaluated by 18F-FDG and 68Ga-FAPI PET/CT in patients with CD.

DETAILED DESCRIPTION:
Patients with intestinal stricture will undergo 18F-FDG and 68Ga-FAPI PET/CT on two consectutive days. The accumulation of 18F-FDG and 68Ga-FAPI at the site of stricture will be determined by standard uptake value (SUV), molecular volume (MV), and total molecular index (TMI). In patients with a planned surgical resection of one or more stricture (s), the image results will be compared with histological findings.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed
* Crohn's disease patients with proofs of intestine stricture by other modalities, e.g. MRI, CT, ultrasound, and/or endoscopy.

Exclusion Criteria:

* Known hypersensitivity to any of the excipients of 18F-FDG and 68Ga-FAPI.
* If the patients are on metformin, discontinuation of 48 hours is required before 18F-FDG injection to minimize the bowel uptake.
* Pregnant or breast-feeding women.
* Any mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study, and/or evidence of an uncooperative attitude.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
SUVmax of stenotic intestine | Day 30 after PET scan
  The SUVmax of stenotic intestine will be determined on 18F-FDG and 68Ga-FAPI PET scan to reflect the highest extent of inflammation and fibrosis, respectively.
MV of stenotic intestine | Day 30 after PET scan
  The MV of stenotic intestine will be determined on 18F-FDG and 68Ga-FAPI PET scan to reflect the involved area of inflammation and fibrosis, respectively.
TMI of stenotic intestine | Day 30 after PET scan
  The TMI of stenotic intestine will be determined on 18F-FDG and 68Ga-FAPI PET scan to reflect the overall extent of inflammation and fibrosis, respectively.

SECONDARY OUTCOMES:
Histological findings | Day 90 after surgery
  In patients with surgical resection of stenotic intestine, the extent of inflammation and fibrosis will be determined.

IPD SHARING:
Plan to Share IPD: Undecided